CLINICAL TRIAL: NCT03952858
Title: Early Telerehabilitation After Hospital Discharge From Acute Care in Geriatric Patients. A Randomized Study With Four, Eight Weeks and Six Months Follow-up
Brief Title: Telerehabilitation in Geriatric Patients at Aarhus University Hospital, Denmark
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Too few elible patients but only one gave informed consent
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Telerehab
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2019-05

CONDITIONS: Frail Elderly Syndrome
Keywords: telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants in the two groups will be asked not to inform the test investigator to which intervention they have been allocated. Baseline test will be performed before randomization in the hospital ward or in the participants home. Before re-test the participants in the intervention groups will ensure that the computer used for exercise is not visible in the room where the re-test is done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): Physiotherapist-supervised Telerehabilitation as home exercise in Groups. Participants in the intervention group receive supervised Telerehabilitation by an experienced physiotherapist two days a week during four weeks. A computer and a camera will be installed where the exercise should take place. It will make it possible for the physiotherapist to see how the participants follow the exercise program and for the participants to follow the physiotherapist instructions on the screen. The participants will be instructed in the use of computer and receive a written guide. After four weeks the participants will on their own continue the Otago exercise Program for another 4 weeks by video sessions and still together in their already established groups. Otago Exercise Program consist of a walking plan, balance exercises, and a set of leg muscle strengthening exercises all progressing in degree of difficulty.
  Interventions: Other: Telerehabilitation Group
- Community Center group (Active Comparator): The Community Center Group will receive the traditional exercise programs offered in a Community Center for older people. The exercise program can vary dependent on the offer in the individual community center. Often the training consists of exercises carried out in a range of different training equipments such as exercise bikes, steppers, rowing machines etc. often supervised by a physiotherapist. At some community centers the training will be performed in groups on appointed times. Some citizens are offered one or two times instruction and hereafter they have to train on their own. Some times the citizens are offered few times of training in their own home and hereafter follow the offer at the community center for older people. Before discharge, at the hospital, their plan for rehabilitation will be completed.
  Participants in the Community Center Group will be tested by the same instruments at baseline and after 4 and 8 weeks and at 6 months of follow-up.
  Interventions: Other: Telerehabilitation Group

INTERVENTIONS:
Other: Telerehabilitation Group — The telerehabilitation Group receives physiotherapy supervised exercises on-line. The Community Center Group receives the traditionel training offer in the municipality Center for older people.
  Other Names: Community Center Group

SUMMARY:
Background Older patients admitted to an Emergency Department (ED) are dependent on assistive devices and almost 16 % have no gait function. It seems appropriate to identify patients who need physical exercises immediately after discharge to avoid further functional decline. New IT technologies make it possible to both supervise the exercises and communicate with the patients via video conferencing equipment. Until now no studies have examined if the Otago Exercise Program (OEP) supervised by video conferencing may enhance motivation and maintain or improve physical functional capacity in acute elderly patients.

Hypothesis Early telerehabilitation performed in groups based on the OEP is compared with traditional exercise programs offered in the community centers in geriatric patients after hospital discharge from acute care.

The study is a randomized, controlled study conducted at Aarhus University Hospital (AUH). The population is elderly patients ≥65 years, residents in the Municipality of Aarhus and admitted acutely from there own home to the ED.

Telerehabilitation Group (TG) will start telerehabilitation first to second week after discharge. After the initial two training sessions, the patient will be included in a TG. When there is a group of two to three participants the group will stop including more members in that group in order to achieve the expected benefits of group exercising. It will be possible for physiotherapists to follow the team on the screen and to communicate with the participants. In addition, the participants may communicate with each other. The following four weeks the patients will exercise on their own in their training groups on appointed times via videoconferencing equipment.

The Control Group will receive the usual training offered by the municipality. Participants in both groups will be tested with the same instruments at baseline and after four and eight weeks and at six months.

Perspective If the presented project indicates that the older target group may benefit from telerehabilitation immediately after discharge, elderly patients may increase their Quality of Life and the municipalities may experience public savings.

Telerehabilitation may be a good alternative for patients who aren't able to receive training at the community center for physical reasons. Telerehabilitation may be one of the means to meet the challenge of the increasing proportion of elderly people in Denmark.

DETAILED DESCRIPTION:
Background The geriatric patient is often presented with a complex pathological picture, where gait- and balance disturbances are independent risk factors for fall accidents, which are common causes for admittance to hospital. One third of the medical patients discharged after an acute hospitalization experience a decrease in functional capacity following one year after. Impaired gait function also greatly influences the older persons' management of their everyday life e.g. transportation, shopping, meals, and domestic tasks. It may induce fear of falling and can lead to isolation and loneliness.

A hip fracture may have fatal consequences. Half of those who are affected of a hip fracture suffer from disabilities, and 15-25% dies within the first year after the trauma.

A program combining exercises of muscle strength, body balance and endurance can break a vicious spiral. Therefore, it seems appropriate to identify those patients who need physical exercises during their hospital stay and immediately after discharge to avoid further functional decline.

Exercise at home and improvement in the ability to undertake daily tasks are highly valued by community-dwelling people 60 years and older. Communication between the older person and the physiotherapist has positive effects on adherence to an exercise program and its outcome.

New Telerehabilitation Technologies make it possible for the physiotherapist to supervise and communicate with exercising participants by video conferencing equipment.

The Otago Exercises Program (OEP) is a home-based strength- and balance program and has proven to reduce falls and injuries caused by fall by 35% in community dwelling older women.

Until now, no studies have examined if OEP supervised through video "face to face" conferencing may maintain or even improve physical functional capacity in older acutely ill patients just discharged to their home. No studies have investigated whether it is possible to carry out Telerehabilitation in groups of geriatric patients aged 65 years or older.

Objective To compare the effect on physical functional capacity by two types of exercises: 1) physiotherapist-supervised Telerehabilitation as home exercise in groups, 2) traditional exercise programs offered in a community center for older people. The target population is 65+ years old home-dwelling medical- and hip fracture patients just discharged after an acute hospitalization.

Hypothesis

Early Telerehabilitation performed in groups based on the Otago exercise program is compared with traditional exercise programs offered in the community centers in geriatric patients after hospital discharge from acute care and supervised by a physiotherapist:

1. Maintain or improve the patient's physical functional abilities within 4 and 8 weeks and 6 months after discharge
2. Prevent loneliness and fear of falling, and maintain or improve the Quality of Life within 4 and 8 weeks and 6 months after discharge Material and methods Design The study is a randomized, controlled parallel-group (two groups), investigator-blinded study.

Population and setting The population is residents living in their own home in the Municipality of Aarhus aged 65 years or older and acutely admitted to Aarhus University Hospital (AUH) in the Emergency Department (ED), and the Departments of Geriatric. The study will be conducted in the community centers for older people, and in the participants' own home.

Participants' recruitment procedure Recruitment will be performed by the project manager in the hospital. All recruitments will be made on weekdays. Eligible patients discharged directly from the ED on weekends or on public holidays will be included on the first weekday after.

Randomization Participants who agree to participate will be randomized to either the Telerehabilitation Group- or the Control Group by a computer-based block randomization via REDCap. It is estimated that it will take about three to four weeks to include three participants in the Intervention Group. It means that the last patient will be included four weeks later than the first included patient. To give the optimal conditions for the home exercise in groups we have in cooperation with the REDCap data manager chosen to modify the randomization from a two block randomization to a three block randomization where two of the blocks allocate participants to the Telerehabilitation Group. Additionally the randomization will stratify the participants according to social status.

Data collection Data will be collected by a skilled test therapist investigator. A gap of plus-minus two days in the re-test follow-up period is accepted.

Sample size calculation To calculate the sample size we use an unpublished study from Hvidovre Hospital (The Capital Region of Denmark). It is older patients who were admitted to the ED that achieved an average score improvement of 1.8 points (SD: 12.8) in the De Morton Mobility Index (DEMMI) after an exercise intervention from admission to four weeks after discharge. DEMMI is a functional test measuring mobility. The Hvidovre study shows that it is necessary to include 27 participants in each group to achieve statistical significance. Likewise, we expect that the participants in our study belong to the same target group as those in the study from Hvidovre, and that their calculation of the sample size also can be applied in our study. It results in a total of 54 participants divided into two identical groups. The study 'Early geriatric follow-up' finds that 16% of community dwelling elderly died within the first 8 weeks after discharge, thus we added another 9 participants i.e. total of 63 participants. Almost 11% will be transferred to a rehabilitation center after discharge (unpublished ref), requiring a total of 70 participants. In an exercise study 22.6 % did not complete their training program, thus it is necessary to include 16 extra participants resulting in a final number of 86 participants i.e. 43 participants in each groups.

Study groups Participants in the Telerehabilitation Group receive supervised Telerehabilitation by an experienced physiotherapist two days a week during four weeks with at least one day of rest between each exercise session (in total: eight Telerehabilitation sessions). Initially the physiotherapist visits the patient at home, and the patient will be informed by a written pamphlet and orally about the exercise program, the benefits of exercise and the expected effect of the program. The patient will be instructed in the use of computer and receives a written guide. New clinical guidelines recommend that geriatric patients should exercise for at least 8 weeks if clinical benefits are to be expected. Therefore, after four weeks the participants will on their own continue OEP for another 4 weeks.

The Telerehabilitation Group will start their exercise within the first week after discharge. When there are a total of two to three participants in the Telerehabilitation Group we will stop including more members in order to achieve the expected benefits of group exercising.

The following four weeks the participants will exercise without supervision by a physiotherapist. The training sessions will continue in their group on appointed times and it will still be possible to communicate with the other participants via computer. Here OEP is displayed on the computer by small video sessions.

The Control Group will receive the usual exercise programs offered in the community center for older people. The exercise program can vary dependent on the offer in the individual community center. Often the training consists of exercises carried out in a range of different training equipment such as exercise bikes, steppers, rowing machines etc. often supervised by a physiotherapist. At some community centers the training will be performed in groups on appointed times. Participants in the Control Group will be tested by the same instruments at baseline and after 4 and 8 weeks and at 6 months of follow-up.

Training intervention OEP consist of a walking plan, balance exercises, and a set of leg muscle strengthening exercises all progressing in degree of difficulty.

The IT platform used in this study make it possible for up to eight persons to see and communicate with each other. We decided because of the heterogeneity among the participants and hereby their different levels of functional capacity to limit the number of participants to three persons joining the intervention group.

In case of cancellation of exercise Participants in both groups who cannot attend the exercise program due to illness, hospitalization or vacation, will remain in their exercise group and finish training on the initially planned date.

Standardization of intervention Before starting the project period, the test investigator will undergo training in performing the tests used in the project to ensure consistency between the testers. The training will be based on the test's appurtenant manuals.

Adherence To achieve the expected effects of the interventions it is crucial that the participants are adherent to the interventions. Therefore the training physiotherapist will register how many times the participants have participated in the training sessions.

In the Control Group, the training physiotherapist in the municipality will be asked to notice how many times participants have received training in the same period. Reasons for non-participation will be noticed in both groups.

Statistical analysis The statistical analysis will be conducted by using STATA (version 15, STATA Corporation, Texas). Baseline data in the Intervention- and Control Group will be compared and presented as means with standard deviations, medians with interquartile ranges or frequencies with percentages depending on data characteristics.

The four time-point FRS mean score will be compared in the two groups in a univariate repeated measurements ANOVA. We assume that the mean-differences are normally distributed, the standard deviations between all time-points are equal, and the differences between all time-point are correlated. We are testing the hypothesis of parallel mean curves with the within and between subject variation between the groups.

Likewise, the four time-points in the DEMMI, and handgrip strength, FES-I, EQ-5 D, GDS and UCLA scores will be tested. A multiple linear regression model is used to analyze if the change in mobility is associated with the change in FES-I, UCLA and EQ-5D in all patients. The model is adjusted for potentially mediating variables: gender, age, social status, comorbidity, educational attainment, and alcohol.

Publication process The results of the study will be presented at relevant internationally conferences. The project manager is employed by Department of Geriatrics as a PhD student in the period of data collection and analysis of data. Department of Geriatrics, Aarhus University Hospital is warrantor of the project.

Ethics The study is approved by the Research Ethics Committee of The Central Denmark Region (1-10-72-394-17) and by the Danish Data Protection Agency (1-16-02-201-17). Participants will be informed that participation is voluntary, they can withdraw at any time without losing their right to treatment. Participants who agree to participate will be requested informed consent. Once written informed consent is obtained from the participants during hospitalization at the ED they will be included in the study. There will be given written and verbal information about the study to ensure that everything is understood and possible questions answered. The Ethic Committee will be informed if important protocol modifications for approval. Communication between patient and therapist will be carried out via the Internet in a secure system.

Blinding It is not possible to blind the participants in relation to the intervention. Also, it is not possible to blind the physiotherapists who are training the participants according to allocation. It is possible, however, to blind the test therapist who will not be advised about to which group the participant is randomized. The primary investigator recruits the participants, screen them for eligibility and collects baseline data before randomization.

Conclusion In a RCT design, the effect of Telerehabilitation within the first week after hospital discharge will be evaluated and compared with the usual training intervention in the municipality in home-dwelling geriatric patients. Change in physical function capacity, loneliness, Quality of Life and fear of falling before and after the interventions are the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* dependent on a walking aid at discharge
* familiar with the use of computer
* informed consent

Exclusion Criteria:

* terminal illness
* inability to walk independent with a walking aid
* inability to speak or understand Danish
* dementia i.e. Short Portable Mental Status Questionnaire (SPMSQ) score above 4
* acute stroke
* inability to complete the Otago Exercise Program without having a great risk of falling

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Instrumental Activities of Daily Living (IADL) | Measured at baseline and after 4 and 8 weeks and after 6 months
  IADL is measured by Functional Recovery Score (FRS). FRS is a questionnaire divided into three subjects such as Basic Activities of Daily Living (BADL), Instrumental Activities of Daily Living (IADL) and mobility (range 0-100 point).

SECONDARY OUTCOMES:
Degree of loneliness | Measured at baseline and after 4 and 8 weeks and after 6 months
  is measured by the University of California Los Angeles Loneliness Scale (UCLA). UCLA is a questionnaire consisting of 20 sub-questions describing subjective feelings of loneliness.
Health-related quality of life and functional ability | Measured at baseline and after 4 and 8 weeks and after 6 months
  measured by European Quality of Life-5 Domain (EQ-5D). It is a generic health-related quality of life instrument that has been used to describe population health and health outcomes in clinical trials. EQ-5D measures quality of life and functional capacity.
Fear of falling | Measured at baseline and after 4 and 8 weeks and after 6 months
  Fear of falling is measured by the Falls Efficacy Scale International (FES-I). FES-I is a questionnaire using a face-to-face interview. It consists of 14 questions.
Mobility | Mobiliy measured by Active Pal is measured after 4 weeks and 6 month
  Mobility is measured by Active Pal. Active Pal is a sensor placed on the thigh. It is able to measure a person's mobility up to seven days. It measures the number of steps and the time the person's femur is placed in both horizontal or vertical position and the number of minutes the person transfers from sitting to a standing position
Balance and mobility | A functional test, which consists of 15 items and measures mobility among frail elderly who are lying in bed or sitting in a comfort chair and the elderly, who are independent in everyday life.
  The De Morton Mobility Index

CONTACTS AND LOCATIONS:
Overall Officials: Bodil K.B. Jørgensen, MHS, Principal Investigator — AUH, Department of Geriatric, Palle Juul-Jensens Bld 8200 Aarhus N, DK; Else marie S. Damsgaard, Professor, Study Chair — AUH, Department of Geriatric, Palle Juul-Jensens Bld. 99, 8200 Aarhus N, Dk; Merete Gregersen, PhD, Study Director — AUH, Department of Geriatric, Palle Juul-Jensens Bld. 99, 8200 Aarhus N, Dk
Locations (2):
- Denmark (2):
  - Department of Geriatric, Aarhus University Hospital, Palle Juul-Jensens Bld. 99, Aarhus
  - Department of Geriatrics, AUH, Aarhus N

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buurman BM, Hoogerduijn JG, de Haan RJ, Abu-Hanna A, Lagaay AM, Verhaar HJ, Schuurmans MJ, Levi M, de Rooij SE. Geriatric conditions in acutely hospitalized older patients: prevalence and one-year survival and functional decline. PLoS One. 2011;6(11):e26951. doi: 10.1371/journal.pone.0026951. Epub 2011 Nov 14. PMID 22110598
- [Background] Ganz DA, Bao Y, Shekelle PG, Rubenstein LZ. Will my patient fall? JAMA. 2007 Jan 3;297(1):77-86. doi: 10.1001/jama.297.1.77. PMID 17200478
- [Background] Mahlknecht P, Kiechl S, Bloem BR, Willeit J, Scherfler C, Gasperi A, Rungger G, Poewe W, Seppi K. Prevalence and burden of gait disorders in elderly men and women aged 60-97 years: a population-based study. PLoS One. 2013 Jul 24;8(7):e69627. doi: 10.1371/journal.pone.0069627. Print 2013. PMID 23894511
- [Background] Lieberman D, Galinsky D, Fried V, Grinshpun Y, Mytlis N, Tylis R. Geriatric Depression Screening Scale (GDS) in patients hospitalized for physical rehabilitation. Int J Geriatr Psychiatry. 1999 Jul;14(7):549-55. doi: 10.1002/(sici)1099-1166(199907)14:73.0.co;2-4. PMID 10440975
- [Background] Wilber ST, Blanda M, Gerson LW. Does functional decline prompt emergency department visits and admission in older patients? Acad Emerg Med. 2006 Jun;13(6):680-2. doi: 10.1197/j.aem.2006.01.006. Epub 2006 Apr 11. PMID 16609104
- [Background] Hoang OT, Jullamate P, Piphatvanitcha N, Rosenberg E. Factors related to fear of falling among community-dwelling older adults. J Clin Nurs. 2017 Jan;26(1-2):68-76. doi: 10.1111/jocn.13337. Epub 2016 Oct 9. PMID 27723217
- [Background] Faulkner KA, Cauley JA, Zmuda JM, Griffin JM, Nevitt MC. Is social integration associated with the risk of falling in older community-dwelling women? J Gerontol A Biol Sci Med Sci. 2003 Oct;58(10):M954-9. doi: 10.1093/gerona/58.10.m954. PMID 14570865
- [Background] Shankar A, McMunn A, Demakakos P, Hamer M, Steptoe A. Social isolation and loneliness: Prospective associations with functional status in older adults. Health Psychol. 2017 Feb;36(2):179-187. doi: 10.1037/hea0000437. Epub 2016 Oct 27. PMID 27786518
- [Background] Nymark T, Lauritsen JM, Ovesen O, Rock ND, Jeune B. Decreasing incidence of hip fracture in the Funen County, Denmark. Acta Orthop. 2006 Feb;77(1):109-13. doi: 10.1080/17453670610045777. PMID 16534709
- [Background] Kjøller M, Davidsen M, Juel K, Sundhedsstyrelsen. Ældrebefolkningens sundhedstilstand i Danmark. Kbh.: Sundhedsstyrelsen
- [Background] Robertson MC, Campbell AJ, Gardner MM, Devlin N. Preventing injuries in older people by preventing falls: a meta-analysis of individual-level data. J Am Geriatr Soc. 2002 May;50(5):905-11. doi: 10.1046/j.1532-5415.2002.50218.x. PMID 12028179
- [Background] Brovold T, Skelton DA, Bergland A. Older adults recently discharged from the hospital: effect of aerobic interval exercise on health-related quality of life, physical fitness, and physical activity. J Am Geriatr Soc. 2013 Sep;61(9):1580-5. doi: 10.1111/jgs.12400. Epub 2013 Aug 8. PMID 23927819
- [Background] Geraedts H, Zijlstra A, Bulstra SK, Stevens M, Zijlstra W. Effects of remote feedback in home-based physical activity interventions for older adults: a systematic review. Patient Educ Couns. 2013 Apr;91(1):14-24. doi: 10.1016/j.pec.2012.10.018. Epub 2012 Nov 26. PMID 23194823
- [Background] World Health Organization. Defining Adherence: section 1 - Setting the scene: chapter one - Defining Adherence. In: World Health Organization, editor. Adherence to Long Term Therapies - Evidence for action
- [Background] Gardner MM, Buchner DM, Robertson MC, Campbell AJ. Practical implementation of an exercise-based falls prevention programme. Age Ageing. 2001 Jan;30(1):77-83. doi: 10.1093/ageing/30.1.77. PMID 11322678
- [Background] Davenport SJ, de Morton NA. Clinimetric properties of the de Morton Mobility Index in healthy, community-dwelling older adults. Arch Phys Med Rehabil. 2011 Jan;92(1):51-8. doi: 10.1016/j.apmr.2010.08.023. PMID 21187205
- [Background] de Morton NA, Davidson M, Keating JL. Validity, responsiveness and the minimal clinically important difference for the de Morton Mobility Index (DEMMI) in an older acute medical population. BMC Geriatr. 2010 Sep 30;10:72. doi: 10.1186/1471-2318-10-72. PMID 20920285
- [Background] Pedersen MM, Petersen J, Bean JF, Damkjaer L, Juul-Larsen HG, Andersen O, Beyer N, Bandholm T. Feasibility of progressive sit-to-stand training among older hospitalized patients. PeerJ. 2015 Dec 17;3:e1500. doi: 10.7717/peerj.1500. eCollection 2015. PMID 26713248
- [Background] Pedersen LH, Gregersen M, Barat I, Damsgaard EM. Early geriatric follow-up after discharge reduces mortality among patients living in their own home
- [Background] Holst M, Sondergaard LN, Bendtsen MD, Andreasen J. Functional training and timed nutrition intervention in infectious medical patients. Eur J Clin Nutr. 2016 Sep;70(9):1039-45. doi: 10.1038/ejcn.2016.72. Epub 2016 Jun 15. PMID 27302668
- [Background] Lord SR, Lloyd DG, Nirui M, Raymond J, Williams P, Stewart RA. The effect of exercise on gait patterns in older women: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 1996 Mar;51(2):M64-70. doi: 10.1093/gerona/51a.2.m64. PMID 8612105
- [Background] Eckardt N. Lower-extremity resistance training on unstable surfaces improves proxies of muscle strength, power and balance in healthy older adults: a randomised control trial. BMC Geriatr. 2016 Nov 24;16(1):191. doi: 10.1186/s12877-016-0366-3. PMID 27881086
- [Background] Ishigaki EY, Ramos LG, Carvalho ES, Lunardi AC. Effectiveness of muscle strengthening and description of protocols for preventing falls in the elderly: a systematic review. Braz J Phys Ther. 2014 Mar-Apr;18(2):111-8. doi: 10.1590/s1413-35552012005000148. Epub 2014 Apr 22. PMID 24760166
- [Background] Smaerup M, Gronvall E, Larsen SB, Laessoe U, Henriksen JJ, Damsgaard EM. Exercise gaming - a motivational approach for older adults with vestibular dysfunction. Disabil Rehabil Assist Technol. 2017 Feb;12(2):137-144. doi: 10.3109/17483107.2015.1104560. Epub 2016 Jan 4. PMID 26727034
- See also: Sundhedsstyrelsen, Statens Institut for Folkesundhed. Danskernes sundhed.dk. 2017 — http://www.danskernessundhed.dk
- See also: Otago Exercise Programme, to prevent falls in older adults — http://www.hret-hiin.org/Resources/falls/16/OtagoExerciseProgramTrainingManualFall2013.pdf
- See also: University V. REDCap — https://redcap.au.dk/
- See also: IT - anvendelse i befolkningen - Danmarks statistik. 2017 — http://www.dst.dk/da/Statistik/Publikationer/VisPub?cid=20739